CLINICAL TRIAL: NCT03317678
Title: Fermented Milk Product With Probiotic and Its Impact on Mood of Patients With Treatment Resistant Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16060902
Record Dates: First submitted 2017-06-06; First posted 2017-10-23 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BioKefir (BKP) (Experimental): BioKefir™ (Lifeway Foods) is a lactose-free fermented milk drink containing 12 different species of bacteria within the lactobacillus, bifidobacterium, and streptococcus generas totaling approximately 20 CFU per 3.5 ounce serving. The product also contains 2 g of fiber, including pectin and inulin. These fibers, especially inulin, are prebiotics that may function along with the probiotic species to support gastrointestinal health. The product is available commercially. Participants will be asked to consume 3.5 ounces twice daily, preferably at morning and nighttime. The probiotic will be provided in individual 3.5 ounce unlabeled containers. These quantities will be started on the first day of the intervention phase of the study (day 0, visit 0) and remain unchanged until the end of the intervention phase on day 56 (visit +4). Administration will be discontinued then.
  Interventions: Dietary Supplement: BioKefir
- Non-fermented Milk (NFM) (Placebo Comparator): The NFM is dairy-based product ultra-filtered to remove lactose. In addition to being matched to lactose, the NFM contains similar energy, fat, and protein content as the probiotic. Participants will be asked to consume 3.5 ounces twice daily, preferably at morning and nighttime. The NFM control will be provided in 11.5 ounce unlabeled containers. These quantities will be started on the first day of the intervention phase of the study (day 0, visit 0) and remain unchanged until the end of the intervention phase on day 56 (visit +4). Administration will be discontinued then.
  Interventions: Dietary Supplement: Non-fermented milk

INTERVENTIONS:
Dietary Supplement: BioKefir — BKP BioKefir (Lifeway Foods) is a lactose-free fermented milk product containing 12 different bacteria provided in a drink.
  Arms: BioKefir (BKP)
Dietary Supplement: Non-fermented milk — A non-fermented milk drink.
  Arms: Non-fermented Milk (NFM)

SUMMARY:
This study aims to assess the impact of a chronic dietary intervention (8 weeks) with probiotics, specifically Fermented Milk Product with Probiotic (FMPP), on the mood of individuals with Major Depressive Disorder (MDD) refractory to standard antidepressant therapy, and its association with changes in intestinal microbiota and markers of inflammation.

DETAILED DESCRIPTION:
Theories about the association of imbalances in the gastro-intestinal (GI) microbiota and its impact on mood states have long existed in medicine. These theories were considered "dead" for most of the 20th century, but converging lines of evidence are now rekindling interest in a link between the GI microbiota and the central nervous system. Newer lines of investigation have made these dormant theories relating commensal microbiota and mood states not only plausible, but the focus of well-designed basic research studies (Yano et al, 2015; Hsiao et al, 2013). The microbial world influence on brain development and behavior was defined by Dr Tom Insel, the former director of the National Institutes of Mental Health as one the "great frontiers" of neuroscience in the next decade (Insel, 2012). Dr. Francis Collins, Director of the National Institutes of Health, further underscored the need for research on the impact of intestinal microbiota on brain function (Collins, 2014).

This renewed interest in understanding the role of the microbiota beyond the digestive tract was spurred in 2007 when the Human Microbiome Project was launched. (Turnbaugh et al, 2007). With over one million different genes and a mass equal to that of the human brain, the genetic diversity of our bacterial commensals outnumbers the human genome by a factor of over 100 to one, and suggests the potential for the genetic variability in the GI environment to impact other body systems, including the central nervous system (CNS). A range of neurotransmitters relevant to mood and anxiety disorders including serotonin, GABA, acetylcholine and endocannabinoids are produced by intestinal microbiota (Dinan et al, 2013). This accruing data along with previous findings showing that pathological gut bacterium are capable of inducing changes in behavior (Lyte et al, 1998) and that early life stress, an established risk factor for major depression, induces changes in the microbiota (O'Mahony et al, 2007) underscore the potential importance of further examining the relationship between the microbiota and brain function with particular attention to the potential therapeutic implications for treatment of psychiatric conditions, such as depression

Preclinical studies demonstrated that noninvasive methods that alter gut microbiota are capable of inducing antidepressant like effects in rat models of depression (Desbonnet et al, 2010). Findings in human populations showed differences in gut flora of depressed individuals when compared to healthy controls, including higher levels of Bacteroidetes, Proteobacteria and Actinobacteria, and a negative correlation between Faecalibacterium and the severity of their depression (Jiang et al, et al 2015). Other studies point to a beneficial effect of probiotics on mood and anxiety in normal volunteers (Messaoudi et al, 2011; Benton et al, 2007), as well as in individuals with Irritable Bowel Syndrome (O' Mahoney et al, 2005) and Chronic Fatigue Syndrome (Rao et al, 2009). However, there have been no systematic studies to date reporting on the impact of probiotics on mood in individuals with major depression.

The majority of depressed patients remain symptomatic despite treatment with currently available antidepressants, and a significant proportion do not respond at all. Thus, the development of new effective antidepressant interventions remains a significant unmet public health need. Given the accumulating evidence for a relationship between the gastrointestinal microbiota and the central nervous system functioning and pathophysiology, including that of affective disorders, it is cogent to measure the impact of probiotic interventions in individuals with refractory depression. The present study proposes to examine the gut microbiota, inflammatory milieu and impact of probiotics on mood in a population of individuals who have been refractory to treatment with standard antidepressant agents.

This study aims to assess the impact of a chronic dietary intervention (8 weeks) with probiotics, specifically Fermented Milk Product with Probiotic (FMPP), on the mood of individuals with Major Depressive Disorder (MDD) refractory to standard antidepressant therapy, and its association with changes in intestinal microbiota and markers of inflammation.

Specific Aim 1. Examine the effect of 8 weeks of probiotic administration on depressive symptoms in depressed patients.

Specific Aim 2. Examine the intestinal microbiota at initiation and end of probiotic administration in order to assess the relationship of baseline and changes in gut flora with treatment response.

Specific Aim 3. Examine baseline and endpoint inflammatory biomarkers including C-reactive protein (CRP) and cytokines to assess the relationship of inflammation with intestinal microbiota and treatment response.

ELIGIBILITY:
Inclusion Criteria

1. Men and women between 21 and 65 years of age meeting DSM-V criteria for Major Depressive Disorder and presenting a HAM-D score of 18 or higher.
2. If patients are on antidepressants (ie. fluoxetine 20 mg/d or its equivalent) the dose needs to be stable for at least 6 weeks prior to screening.
3. Patients with Body Mass Indexes between 18 and 40.
4. No planned antibiotic treatment during study to avoid antibiotic treatments for the duration of the study.

Exclusion Criteria

1. Patients who are vegan or observe other specific dietary patterns that are not representative of the general population and may specifically impact their microbiomes will be excluded from the study.
2. Lactose intolerant patients will not be able to participate due to the high likelihood of being unable to tolerate the specific intervention being implemented.
3. Patients who have used BKP or Yogurt without probiotics daily for 12 weeks preceding study entry and unwilling to stop.
4. Patients with a past history of Eating Disorders or Psychotic Disorders. Patients with Bipolar Disorder, past or current, who are currently taking a mood stabilizer.
5. Patients with Substance Use Disorder. Within the past 12 months.
6. Patients with a history of 3 or more failed trials of antidepressant medications of adequate dose or duration (i.e. fluoxetine 20 mg/d or its equivalent for 6 weeks or more).
7. Patients with other significant clinical illnesses such as, but not limited to, Congestive Heart Failure, Diabetes Mellitus, Chronic Obstructive Pulmonary Disease.
8. Patients who are currently using corticosteroid medications, or who have a history of multiple treatment courses with these medications.
9. Patients on antibiotic treatment at the time of study entry or who have received such treatment during the 30 days prior to study entry.
10. Patients using anti-inflammatory medications.
11. Patients who are actively suicidal.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Changes in total score on the Montgomery-Åsberg Depression Rating | Baseline assessments and every 2 weeks over 91 days
  The primary outcome measure will be change in the Montgomery-Åsberg Depression Rating Scale (MADRS). The MADRS is a 10-item scale for the evaluation of depressive symptoms (Montgomery & Åsberg, 1979).

SECONDARY OUTCOMES:
Changes in Clinical Global Impression-Severity Scale (CGI) | Baseline assessments and every 2 weeks over 91 days
  Change in the Clinical Global Impression-Severity Scale (CGI) from baseline to weekly assessments. The CGI is a 7 point scale that measures symptom illness and global improvement or changes in severity
Change in total score on the Computerized Adaptive Testing for Depression (CAT-D) | Baseline assessments and every 2 weeks over 91 days
  CAT-D is a multidimensional item response questionnaire that selects a small-targeted set of items for each individual from a much larger bank of test items. CAT yields scores ranging from 0 to 100 and these will be used to assess changes in participants' mood from baseline and weekly assessments.
Analysis of Intestinal Microbiota pre and post intervention | Baseline and after 56 days of intervention.
  A quantitative analysis of the fecal microbiome will be conducted

CONTACTS AND LOCATIONS:
Locations (1):
- RushUMC, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No